CLINICAL TRIAL: NCT00908739
Title: Assessment of Patterns of Expression of VEGF, Matrix Metalloproteinase 2, 9 Activity, E-Cadherin Regulation and CA-9 Activity as Predictors of Aggressive Renal Cell Carcinoma Behavior
Brief Title: Studying Tumor Tissue Samples From Patients Who Have Undergone Surgery for Localized Kidney Cancer
Status: Withdrawn | Type: Observational
Why Stopped: PI left
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: David A. Levy, Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center
Other Study IDs: CASE1808; P30CA043703 (NIH); CASE1808 (Other: Case Comprehensive Cancer Center); CASE-1808-CC503
Record Dates: First submitted 2009-05-23; First posted 2009-05-27 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage III renal cell cancer; recurrent renal cell cancer; clear cell renal cell carcinoma; childhood renal cell carcinoma
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Gene Expression Profiling; Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Previously collected tumor tissue samples are examined by immunohistochemistry for levels of expression of five different factors related to aggressive tumor behavior (i.e., VEGF expression, E-cadherin regulation, matrix metalloproteinase 2 and 9 activity, and carbonic anhydrase 9 activity.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: gene expression analysis — immunohistochemistry for levels of expression of five different factors related to aggressive tumor behavior (i.e., VEGF expression, E-cadherin regulation, matrix metalloproteinase 2 and 9 activity, and carbonic anhydrase 9 activity)
Other: immunohistochemistry staining method — immunohistochemistry for levels of expression of five different factors related to aggressive tumor behavior (i.e., VEGF expression, E-cadherin regulation, matrix metalloproteinase 2 and 9 activity, and carbonic anhydrase 9 activity)
Other: laboratory biomarker analysis — immunohistochemistry for levels of expression of five different factors related to aggressive tumor behavior (i.e., VEGF expression, E-cadherin regulation, matrix metalloproteinase 2 and 9 activity, and carbonic anhydrase 9 activity)

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor tissue samples from patients who have undergone surgery for localized kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify consistent patterns of VEGF expression, E-cadherin regulation, matrix metalloproteinase 2 and 9 activity, and carbonic anhydrase 9 activity as predictive factors in the development of aggressive tumor behavior in tumor tissue samples from patients with localized clear cell renal cell carcinoma.

OUTLINE: Previously collected tumor tissue samples are examined by immunohistochemistry for levels of expression of five different factors related to aggressive tumor behavior (i.e., VEGF expression, E-cadherin regulation, matrix metalloproteinase 2 and 9 activity, and carbonic anhydrase 9 activity). Samples are compared to positive tissue controls (i.e., VEGF- tonsil; E- cadherin-normal breast or endometrium; MMP2- placenta) and a negative control (i.e., isotype matched normal serum) to identify consistent patterns of expression/activity of these factors. Levels of expression are quantified as 5-level scores (0 to 4 scale) and differences between any two areas of a tumor are analyzed.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Tumor tissue samples from patients who recently underwent nephrectomy or partial nephrectomy for clear cell renal cell carcinoma

  * Harvested from the superior, inferior, left lateral, right lateral, and central portions of resected or discarded tumor measuring 4 cm or less
  * Localized disease (pT1a, N0-Nx, M0)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Relative patterns of expression/activity of five different growth factors/enzymes inherently related to the development of metastatic renal cell carcinoma behavior

CONTACTS AND LOCATIONS:
Overall Officials: David A. Levy, MD, Principal Investigator — Ireland Cancer Center at University Hospitals Case Medical Center, Case Comprehensive Cancer Center